CLINICAL TRIAL: NCT01709825
Title: The Effect of Probiotics on Immune Function, and Digestive Health in Academically-stressed University Students: A Randomized, Double-blinded, Placebo-controlled Study
Brief Title: The Effect of Probiotics (L. Helveticus, B. Longum, and B. Bifidum) on Immune Function and Digestive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Human Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 403-2012
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: probiotics; cold; flu; immune function; microbiota
MeSH Terms: conditions — Common Cold; Influenza, Human | interventions — Sugars; Sucrose; ISL2 protein, Lactobacillus helveticus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sugar Pill (Placebo Comparator): Sugar Pill will be taken as a capsule once daily for 6 weeks.
  Interventions: Dietary Supplement: Sugar Pill
- Probiotic- Bifidobacterium bifidum (Experimental): Bifidobacterium bifidum (Supplement A) will be taken as a capsule once daily for 6 weeks.
  Interventions: Dietary Supplement: Probiotic- Bifidobacterium Bifidum
- Probiotic- Lactobacillus helveticus (Experimental): Lactobacillus helveticus (Supplement B) will be taken as a capsule once daily for 6 weeks.
  Interventions: Dietary Supplement: Probiotic- Lactobacillus helveticus
- Probiotic- Bifidobacterium longum ss. Infantis R0033 (Experimental): Bifidobacterium longum ss. Infantis R0033 (Supplement C)will be taken as a capsule once daily for 6 weeks.
  Interventions: Dietary Supplement: Probiotic- Bifidobacterium longum ss. Infantis R0033

INTERVENTIONS:
Dietary Supplement: Probiotic- Bifidobacterium Bifidum — Bifidobacterium bifidum R0071 will be taken as a capsule once daily for 6 weeks.
  Other Names: Bifidobacterium bifidum; Supplement A
  Arms: Probiotic- Bifidobacterium bifidum
Dietary Supplement: Sugar Pill — Sugar Pill (Sucrose) will be taken as a capsule once daily for 6 weeks.
  Other Names: Sucrose
  Arms: Sugar Pill
Dietary Supplement: Probiotic- Lactobacillus helveticus — Lactobacillus helveticus R0052 will be taken as a capsule once daily for 6 weeks.
  Other Names: Lactobacillus helveticus; Supplement B
  Arms: Probiotic- Lactobacillus helveticus
Dietary Supplement: Probiotic- Bifidobacterium longum ss. Infantis R0033 — Bifidobacterium longum ss. Infantis R0033 (Supplement C) will be taken as a capsule once daily for 6 weeks.
  Other Names: Bifidobacterium longum ss. Infantis R0033; Supplement C
  Arms: Probiotic- Bifidobacterium longum ss. Infantis R0033

SUMMARY:
The purpose of this study is to determine if daily consumption of a probiotic in the period before, during and after academic exams will help maintain digestive and immune health and quality of life of undergraduate students.

DETAILED DESCRIPTION:
A randomized, double-blinded, placebo-controlled trial will be used. Healthy full-time undergraduate students will be recruited from the University of Florida via flyers, emails, announcements, etc. Informed consent will be obtained and the inclusion/exclusion criteria will be reviewed to determine whether a participant qualifies for the study. All participants will be consented for the main six-week intervention and a subgroup (n=50/group) of these students will be consented to provide two stool samples.

Participants will provide saliva and stool samples (for the sub-group)during the pre-baseline week and during the week of final exams at approximately week 4. At the randomization visit, height, weight and age will be obtained. Participants will be stratified based on body mass index and randomized via sealed envelopes to one of four groups: Lactobacillus helveticus, Bifidobacterium longum ssp. Infantis, Bifidobacterium bifidum or the placebo (n=145/group). Participants will take the study provided capsule of probiotic or placebo daily for 6 weeks. Participants will receive daily questionnaires via email throughout the prebaseline week and the 6-week intervention. Daily questionnaires will ask about intake of the supplement, cold symptoms, and general health (i.e., new medications, doctor visits). Throughout the study, participants will also be asked to complete weekly questionnaires (inquiring about gastrointestinal symptoms and physical activity) and Quality of Life Questionnaires (administered during pre-baseline, final exam week and week 6 of the study).

ELIGIBILITY:
Inclusion Criteria:

To participate in the study you must:

* be 18 years of age or older.
* be a healthy full-time undergraduate at the University of Florida.
* be willing to complete daily questionnaires form via computer.
* be willing to discontinue any immune-enhancing dietary supplements (e.g., prebiotics and fiber supplements, probiotics, echinacea, fish oil, vitamin E >400% of the RDA or >60 mg/day).
* be willing to take the probiotic capsule daily of 6 weeks.
* have had at least one cold in the last 12 months.
* have at least 1 final during the scheduled exam week.
* have daily access to the Internet.

Exclusion Criteria:

To participate in the study you must NOT:

* be a current smoker.
* have chronic allergies involving the upper respiratory tract.
* have had immunosuppressive illness or treatment within the last year.
* have received antibiotic therapy in the past two months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of days without cold/flu | over 6 weeks
  The intensity of cold/flu symptoms (running/congested nose, stiffness or chills, headache, cough, fatigue, fever, sore throat, achiness, and ear discomfort)will be scored as 0 (not experiencing) to 3 (severe). The symptom intensity from the 9 cold/flu symptoms will be summed to obtain a symptom intensity score. A symptom intensity score of >6 will be designated as a day of cold. The mean proportion of days without a cold/flu will be compared between each probiotic and the placebo.
Microbiota Study | Change in microbiota from pre-baseline to on average week 4
  * Microbial diversity measured by DGGE profiling (detect large distortions)
  * qPCR to quantify treatment effects on specific bacteria
Digestive Health | Daily for 7 weeks
  * Gastrointestinal symptoms (gas, bloating, diarrhea, etc.)
  * Bowel habits (bowel movement frequency and consistency)
  * Measures of quality of life (physical functioning, general health, bodily pain, vitality and social functioning)

SECONDARY OUTCOMES:
Immune Health | Measured at pre-baseline and on average week 4
  * Salivary secretory immunoglobulin A (sIgA)
  * Fecal sIgA

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida; Wendy Dahl, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Langkamp-Henken B, Rowe CC, Ford AL, Christman MC, Nieves C Jr, Khouri L, Specht GJ, Girard SA, Spaiser SJ, Dahl WJ. Bifidobacterium bifidum R0071 results in a greater proportion of healthy days and a lower percentage of academically stressed students reporting a day of cold/flu: a randomised, double-blind, placebo-controlled study. Br J Nutr. 2015 Feb 14;113(3):426-34. doi: 10.1017/S0007114514003997. Epub 2015 Jan 21. PMID 25604727
- [Derived] Culpepper T, Christman MC, Nieves C Jr, Specht GJ, Rowe CC, Spaiser SJ, Ford AL, Dahl WJ, Girard SA, Langkamp-Henken B. Bifidobacterium bifidum R0071 decreases stress-associated diarrhoea-related symptoms and self-reported stress: a secondary analysis of a randomised trial. Benef Microbes. 2016 Jun;7(3):327-36. doi: 10.3920/BM2015.0156. Epub 2016 Feb 3. PMID 26839075